CLINICAL TRIAL: NCT01686061
Title: Blepharospasm Patient Survey: A Structured Interview Evaluating Previous and Current incobotulinumtoxinA, abobotulinumtoxinA and onabotulinumtoxinA Treatment for Patients With Blepharospasm
Brief Title: Blepharospasm Patient Survey for Patients With Blepharospasm
Status: Completed | Type: Observational
Sponsor: Merz Pharmaceuticals GmbH (Industry)
Collaborators: Merz North America, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: MUS6020100920
Record Dates: First submitted 2012-09-12; First posted 2012-09-17 (Estimated); Last update posted 2022-10-28 (Actual); Status verified 2014-04

CONDITIONS: Blepharospasm
MeSH Terms: conditions — Blepharospasm

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Blepharospasm Survey Group
  Interventions: Other: No intervention- only one time survey

INTERVENTIONS:
Other: No intervention- only one time survey

SUMMARY:
The purpose of this survey is to collect detailed information on patients treated for blepharospasm with incobotulinumtoxinA, abobotulinumtoxinA and onabotulinumtoxinA, including how often they are treated with botulinum toxin, how long their treatment lasts, how satisfied they are with their treatment, and if there is any improvement in their symptoms with the treatment.

DETAILED DESCRIPTION:
This study is open to males and females > 18 years and < 81 years with a clinical diagnosis of blepharospasm.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subject aged > 18 years and < 81 years
* Documented clinical diagnosis of blepharospasm
* Currently receiving incobotulinumtoxinA, abobotulinumtoxinA or onabotulinumtoxinA

Exclusion Criteria:

* Previous treatment with rimabotulinumtoxinB in the last 2 treatment cycles

Ages: 18 Years to 81 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated for blepharospasm with incobotulinumtoxinA, abobotulinumtoxinA or onabotulinumtoxinA treatment.
Sampling Method: Non-Probability Sample
Enrollment: 124 (Actual)
Dates: Start 2012-09; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Botulinum Toxin Treatment Information | This is a single, structured interview about experiences with Botulinum Toxins
  The following information for patients treated for blepharospasm with incobotulinumtoxinA, abobotulinumtoxinA, or onabotulinumtoxinA treatment is collected: (1) botulinum treatment information such as intervals for botulinum injections, physician's rationale for injection interval, overall experience with botulinum toxin injections (onset, maximum effect, decline of effect), current injection cycle experience (current satisfaction, satisfaction at maximum effect, and visual analog scale (VAS) of current health status); and (2) disability status using the Blepharospasm Disability Index (BSDI) and the Jankovic Rating Scale (JRS)

CONTACTS AND LOCATIONS:
Overall Officials: Micki Seoane, Study Director — Merz Pharmaceutical, LLC
Locations (5):
- United States (5):
  - Merz Investigative Site #0007, Fountain Valley, California
  - Merz Investigative Site # 0002, Sarasota, Florida
  - Merz Investigative Site # 0001, Boston, Massachusetts
  - Merz Investigative Site #003, Durham, North Carolina
  - Merz Investigative Site # 0006, Columbus, Ohio